CLINICAL TRIAL: NCT02706925
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses of BI 443651 in Healthy Male Volunteers in a Partially Randomised, Single Blind, Placebo-controlled Trial
Brief Title: To Assess Safety, Tolerability and Pharmacokinetics of BI 443651 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1363.1; 2015-004395-30 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- BI 443651 (Experimental)
  Interventions: Drug: BI 443651
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 443651
  Arms: BI 443651
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability and pharmacokinetics, following single doses of BI 443651

ELIGIBILITY:
Inclusion criteria:

* Healthy male according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* The subject has a diagnosis history of pulmonary hyperreactivity.
* Estimated glomerular filtration rate (eGFR) below 80 mL/min

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2016-06-12 (Actual); Study Completion 2016-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed as a partially randomised, placebo-controlled within parallel dose groups, single-blind trial.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- Placebo: Subjects were administered single dose of matching placebo to BI 443651 solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 10 μg: Subjects were administered single dose of BI 443651 10 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 30 μg: Subjects were administered single dose of BI 443651 30 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 100 μg: Subjects were administered single dose of BI 443651 100 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 300 μg: Subjects were administered single dose of BI 443651 300 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 900 μg: Subjects were administered single dose of BI 443651 900 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 1800 μg: Subjects were administered single dose of BI 443651 1800 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 2700 μg: Subjects were administered single dose of BI 443651 2700 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
- BI 443651 3600 μg: Subjects were administered single dose of BI 443651 3600 μg solution for inhalation per actuation via the RESPIMAT® inhaler orally.
Period: Overall Study
Arm/Group | Placebo | BI 443651 10 μg | BI 443651 30 μg | BI 443651 100 μg | BI 443651 300 μg | BI 443651 900 μg | BI 443651 1800 μg | BI 443651 2700 μg | BI 443651 3600 μg
Started | 16 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Completed | 16 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set includes all subjects from the Randomised Set [(RS: all subjects who entered the trial, i.e., who have been assigned a subject number)] who were documented to have taken at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 443651 10 μg | BI 443651 30 μg | BI 443651 100 μg | BI 443651 300 μg | BI 443651 900 μg | BI 443651 1800 μg | BI 443651 2700 μg | BI 443651 3600 μg | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (9.3) | 31.0 (7.5) | 40.5 (7.2) | 26.8 (1.9) | 30.3 (5.1) | 37.6 (8.3) | 31.5 (7.8) | 31.7 (10.0) | 31.8 (9.7) | 32.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 16 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events (AEs)
Description: This outcome measure presents percentage of the subjects with drug-related AEs. The doses ranged from 10 μg to 3600 μg for the outcome measure [Percentage of subjects with drug-related Adverse Events (AEs)].
Time Frame: Up to 216 hours.
Population: Treated Set (TS): This subject set includes all subjects from the Randomised Set (RS) who were documented to have taken at least 1 dose of study drug.
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo | BI 443651 10 μg | BI 443651 30 μg | BI 443651 100 μg | BI 443651 300 μg | BI 443651 900 μg | BI 443651 1800 μg | BI 443651 2700 μg | BI 443651 3600 μg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Percentage of subjects | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 16.7 | 66.7 | 66.7

2. Secondary Outcome: AUC0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point)
Description: This outcome measure presents area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz).
  Time frame note: The time points 72:00h, 96:00h below was only applicable for highest dose (and corresponding placebo subjects).
  Two blood sample for stability testing were taken at 3:00h time point from the Treatment C dose group only.
  The doses ranged from 10 μg to 3600 μg for the outcome measure [AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)].
Time Frame: 1.30 (hours: minutes) hours (h) before drug administration and 0:05h, 0:10h, 0:15h, 0:20h, 0:30h, 0:40h, 0:50h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h, 72:00h, 96:00h after drug administration.
Population: Pharmacokinetic Analysis Set (PKS): This subject set includes all subjects from the TS on who received Boehringer Ingelheim (BI) 443651 and who provided at least 1 PK endpoint value that was judged as PK evaluable and not affected by protocol violations relevant to the evaluation of PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | BI 443651 10 μg | BI 443651 30 μg | BI 443651 100 μg | BI 443651 300 μg | BI 443651 900 μg | BI 443651 1800 μg | BI 443651 2700 μg | BI 443651 3600 μg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
pmol*h/L | 24.2 (54.7) | 146 (69.4) | 506 (42.5) | 1860 (54.8) | 5680 (57.3) | 26400 (49.8) | 39300 (34.3) | 60700 (43.9)
Statistical Analysis 1: Comparison: BI 443651 10 μg vs BI 443651 30 μg vs BI 443651 100 μg vs BI 443651 300 μg vs BI 443651 900 μg vs BI 443651 1800 μg vs BI 443651 2700 μg vs BI 443651 3600 μg; Test type: Superiority or Other; Slope = 1.2951, 95% CI 2-sided [1.2242 to 1.3660], Standard Deviation 0.0352 — The model of dose proportionality was power model that describes the functional relationship between the dose and PK endpoints. Perfect dose proportionality would correspond to a slope of 1. Standard deviation is actually the standard error of slope
Statistical Analysis 2: Comparison: BI 443651 30 μg vs BI 443651 100 μg vs BI 443651 300 μg vs BI 443651 900 μg; Test type: Superiority or Other; Slope = 1.0880, 95% CI 2-sided [0.9128 to 1.2633], Standard Deviation 0.0843 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BI 443651 1800 μg vs BI 443651 2700 μg vs BI 443651 3600 μg; Test type: Superiority or Other; Slope = 1.1846, 95% CI 2-sided [0.4791 to 1.8900], Standard Deviation 0.3328 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma)
Description: This outcome measure presents maximum concentration of analyte in plasma (Cmax).
  Time frame note: The time points 72:00h, 96:00h below was only applicable for highest dose (and corresponding placebo subjects).
  Two blood sample for stability testing were taken at 3:00h time point from the Treatment C dose group only.
  The doses ranged from 10 μg to 3600 μg for the outcome measure [Cmax (maximum measured concentration of the analyte in plasma)].
Time Frame: as for outcome 2
Population: Pharmacokinetic Analysis Set (PKS): This subject set includes all subjects from the TS on who received BI 443651 and who provided at least 1 PK endpoint value that was judged as PK evaluable and not affected by protocol violations relevant to the evaluation of PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | BI 443651 10 μg | BI 443651 30 μg | BI 443651 100 μg | BI 443651 300 μg | BI 443651 900 μg | BI 443651 1800 μg | BI 443651 2700 μg | BI 443651 3600 μg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
pmol/L | 14.1 (20.7) | 58.7 (81.6) | 198 (35.5) | 725 (41.1) | 1700 (43.0) | 7590 (60.2) | 14400 (39.2) | 19800 (56.2)
Statistical Analysis 1: Comparison: BI 443651 10 μg vs BI 443651 30 μg vs BI 443651 100 μg vs BI 443651 300 μg vs BI 443651 900 μg vs BI 443651 1800 μg vs BI 443651 2700 μg vs BI 443651 3600 μg; Test type: Superiority or Other; Slope = 1.2114, 95% CI 2-sided [1.1409 to 1.2818], Standard Deviation 0.0350 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 443651 10 μg vs BI 443651 30 μg vs BI 443651 100 μg vs BI 443651 300 μg vs BI 443651 900 μg; Test type: Superiority or Other; Slope = 1.0771, 95% CI 2-sided [0.9696 to 1.1845], Standard Deviation 0.0524 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BI 443651 1800 μg vs BI 443651 2700 μg vs BI 443651 3600 μg; Test type: Superiority or Other; Slope = 1.3969, 95% CI 2-sided [0.5563 to 2.2375], Standard Deviation 0.3965 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 1 day after last drug administration, up to 70 days.
Arm/Group | Placebo | BI 443651 10 μg | BI 443651 30 μg | BI 443651 100 μg | BI 443651 300 μg | BI 443651 900 μg | BI 443651 1800 μg | BI 443651 2700 μg | BI 443651 3600 μg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/16 | 1/6 | 0/6 | 0/6 | 2/6 | 2/5 | 3/6 | 4/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | BI 443651 10 μg (N=6) | BI 443651 30 μg (N=6) | BI 443651 100 μg (N=6) | BI 443651 300 μg (N=6) | BI 443651 900 μg (N=5) | BI 443651 1800 μg (N=6) | BI 443651 2700 μg (N=6) | BI 443651 3600 μg (N=6)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No